CLINICAL TRIAL: NCT02935322
Title: Interaction Chlorhexidine-fluoride - a 4-day and 6-week Randomised Clinical Mouthrinse Study
Brief Title: Interaction Between Chlorhexidine and Fluoride
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Oscar Villa, PhD, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dnr 745-11
Record Dates: First submitted 2016-10-10; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Periodontal Disease; Dental Caries
Keywords: Prevention
MeSH Terms: conditions — Periodontal Diseases; Dental Caries | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.12 % chlorhexidine + 0.2 % NaF mouthrinse (Active Comparator): A mouthrinse combining chlorhexidine and NaF
  Interventions: Drug: 0.12 % chlorhexidine + 0.2 % NaF mouthrinse
- 0.2 % NaF mouthrinse (Active Comparator): A mouthrinse containing NaF
  Interventions: Drug: 0.2 % NaF mouthrinse
- 0.12% chlorhexidine mouthrinse (Active Comparator): A mouthrinse containing chlorhexidine
  Interventions: Drug: 0.12% chlorhexidine
- Placebo mouthrinse (Placebo Comparator): A mouthrinse containing all basic ingredients as the other three mouth rinses compared but without chlorhexidine and fluoride
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 0.12 % chlorhexidine + 0.2 % NaF mouthrinse — In study I, subjects were asked to refrain from tooth brushing and interdental cleaning and rinse with 10 ml of the assigned test solution for one minute, twice daily (morning and evening) during 4 days.
  In study II, subjects were asked to rinse with 10ml of the assigned test solution twice daily after tooth brushing during a 6-week period.
  Other Names: Chlorhexidine + NaF mouthwash
  Arms: 0.12 % chlorhexidine + 0.2 % NaF mouthrinse
Drug: 0.2 % NaF mouthrinse — In study I, subjects were asked to refrain from tooth brushing and interdental cleaning and rinse with 10 ml of the assigned test solution for one minute, twice daily (morning and evening) during 4 days.
  In study II, subjects were asked to rinse with 10ml of the assigned test solution twice daily after tooth brushing during a 6-week period.
  Other Names: NaF mouthwash
  Arms: 0.2 % NaF mouthrinse
Drug: 0.12% chlorhexidine — In study I, subjects were asked to refrain from tooth brushing and interdental cleaning and rinse with 10 ml of the assigned test solution for one minute, twice daily (morning and evening) during 4 days.
  In study II, subjects were asked to rinse with 10ml of the assigned test solution twice daily after tooth brushing during a 6-week period.
  Other Names: Chlorhexidine mouthwash
  Arms: 0.12% chlorhexidine mouthrinse
Other: Placebo — Contained all basic ingredients as the other three mouthrinses but no chlorhexidine and no NaF. In study I, subjects were asked to refrain from tooth brushing and interdental cleaning and rinse with 10 ml of the assigned test solution for one minute, twice daily (morning and evening) during 4 days.
  In study II, subjects were asked to rinse with 10ml of the assigned solution twice daily after tooth brushing during a 6-week period.
  Arms: Placebo mouthrinse

SUMMARY:
The aim of the present study was to study if there are interactions and reduced clinical effect between chlorhexidine and fluoride when they are combined in the same mouthrinse.

DETAILED DESCRIPTION:
The investigation assessed the clinical effect of a mouthrinse containing chlorhexidine (CHX) and sodium fluoride (NaF) during a 4-day period of non-brushing and a 6-week period of brushing. Two studies were designed as double-blind, randomized, cross-over clinical trials. In study I, 16 healthy subjects rinsed twice daily for 1 min during 4 days of no tooth brushing with four mouthrinse solutions: 1) 0.12% CHX + 0.2% NaF, 2) 0.2% NaF, 3) 0.12% CHX, and 4) placebo. In study 2, 16 healthy subjects rinsed with the same four solutions twice daily after tooth brushing during a 6-week period. Primary outcomes were plaque formation and gingivitis. Secondary outcomes were fluoride retention and microbiological parameters in plaque and saliva (total bacterial counts and mutans streptococci, lactobacilli and streptococci sanguinis counts). One way analyses of variance with post hoc Student-Newman-Keul´s statistical test was performed for comparisons between mouthrinses. Intragroup changes over time were analyzed with a paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 18-35 years
* Good general health
* No signs of periodontitis and caries
* A minimum of 24 teeth with no extensive restorations
* No current or planned dental treatment during the trial periods.

Exclusion Criteria:

* Antibiotic treatment within 1 month prior to the start of the trial
* Current medication with anti-inflammatory drugs
* Use of antiseptic mouthrinses
* Smokers and snuff user
* Use of chewing gums

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Plaque index | Baseline
Plaque index | Day 4
Plaque index | Day 42
Gingivitis index | Baseline
Gingivitis index | Day 42

SECONDARY OUTCOMES:
Mutans streptococci counts in dental plaque and saliva | Day 0
Mutans streptococci counts in dental plaque and saliva | Day 4
Streptococcus sanguis counts in dental plaque and saliva | Day 42
Lactobacilli counts in dental plaque and saliva | Day 0
Lactobacilli counts in dental plaque and saliva | Day 4
Lactobacilli counts in dental plaque and saliva | Day 42
Streptococcus sanguinis counts in dental plaque and saliva | Day 0
Streptococcus sanguinis counts in dental plaque and saliva | Day 4
Streptococcus sanguinis counts in dental plaque and saliva | Day 42
Total bacterial counts in dental plaque and saliva | Day 0
Total bacterial counts in dental plaque and saliva | Day 4
Total bacterial counts in dental plaque and saliva | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Per Ramberg, Professor, Study Chair — Göteborg University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Axelsson P, Lindhe J. The effect of a preventive programme on dental plaque, gingivitis and caries in schoolchildren. Results after one and two years. J Clin Periodontol. 1974;1(2):126-38. doi: 10.1111/j.1600-051x.1974.tb01248.x. No abstract available. PMID 4532119
- [Background] Barkvoll P, Rolla G, Bellagamba S. Interaction between chlorhexidine digluconate and sodium monofluorophosphate in vitro. Scand J Dent Res. 1988 Feb;96(1):30-3. doi: 10.1111/j.1600-0722.1988.tb01404.x. PMID 3422503
- [Background] Emilson CG. Susceptibility of various microorganisms to chlorhexidine. Scand J Dent Res. 1977 May;85(4):255-65. doi: 10.1111/j.1600-0722.1977.tb00561.x. PMID 266752
- [Background] Dahlen G. Effect of antimicrobial mouthrinses on salivary microflora in healthy subjects. Scand J Dent Res. 1984 Feb;92(1):38-42. PMID 6585909
- [Background] Dolles OK, Bonesvoll P, Gamst ON, Gjermo P. Determination of fluoride and chlorhexidine from chlorhexidine/fluoride-containing dentifrices. Scand J Dent Res. 1979 Apr;87(2):115-22. doi: 10.1111/j.1600-0722.1979.tb00662.x. PMID 292158